CLINICAL TRIAL: NCT05133102
Title: Repeated Sampling of the Oral Microbiome to Improve Detection of Barrett's Esophagus
Brief Title: Longitudinal Oral Microbiome Sampling for BE
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of Michigan (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julian A Abrams, MD, Associate Professor of Medicine and Epidemiology, Columbia University
Other Study IDs: AAAS2622; R01CA238433 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Barrett Esophagus
Keywords: Saliva; Sampling; Oral Microbiome
MeSH Terms: conditions — Barrett Esophagus | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Patients who have undergone an endoscopy within the last three years and have never been diagnosed with Barrett's esophagus.
  Interventions: Other: Sample collection
- Barrett's Esophagus: Patients who have undergone an endoscopy within the last three years and have histologically confirmed Barrett's esophagus. BE segment must be M>1cm, and has not be treated with endoscopic eradication therapy (focal mucosal resection without subsequent eradication therapy is allowed).
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Collection of saliva sample

SUMMARY:
This is a longitudinal cohort study to assess the impact of repeated sampling of an oral microbiome signature for Barrett's esophagus (BE). Potential participants will be identified through chart review of patients who have had an endoscopy in the past three years.

DETAILED DESCRIPTION:
Saliva collection is non-invasive and can be performed in clinical and non-clinical settings. As such, saliva testing is a highly attractive method for diagnosing and/or monitoring disease. The investigators previously showed that the bacterial make-up ("microbiome") of saliva is highly distinct in patients with and without Barrett's esophagus (BE), a precursor to esophageal cancer that normally can only be diagnosed by undergoing an upper endoscopy. While the microbiome of saliva is felt to be relatively stable over time, it is unclear whether a microbiome signature for Barrett's esophagus is reproducible within individuals. Also, repeated testing of saliva may improve the ability to diagnose Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an upper endoscopy or had upper endoscopy within past three years
* Eighteen years of age or older
* Capable of producing a saliva sample
* Able to give informed consent
* For BE patients only: Endoscopic evidence of Barrett's esophagus (at least 1 cm maximal BE length; i.e. Prague classification: any C, M≥1), and intestinal metaplasia present on esophageal biopsies

Exclusion Criteria:

* History of head and neck cancer or esophageal squamous cell or gastric cancer
* History of esophageal or gastric surgery
* Scheduled to undergo colonoscopy on the day of initial saliva collection
* Scheduled only for Endoscopic retrograde cholangiopancreatography (ERCP) or Endoscopy ultrasound (EUS) without accompanying standard upper endoscopy on the day of initial saliva collection
* For BE patients only: History of prior endoscopic therapy for BE except a history of prior Endoscopic mucosal resection (EMR) of focal lesions without subsequent ablative therapy is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment will continue until a total of 250 subjects complete all three saliva specimen collections:
  * 50 BE patients
  * 200 controls
  The investigators anticipate that approximately 10% of subjects will not complete all three specimen collections and will be excluded from the primary outcome analyses. Thus, the investigators expect to enroll ~275 subjects to have 250 with three saliva specimen collections. There is no cap on enrollment per study site. The anticipated duration of enrollment is 2 years (24 months).
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics of a microbiome-based classifier with repeated sampling | 2 months
  Using a classifier developed from 16S rRNA gene sequencing data, the investigators will calculate the area under the receiver operating curve (AUROC) and associated 95% confidence interval for a classifier with three repeated measures per subject.
Intra-class correlation coefficients (ICC) by BE status | 2 months
  This will be measured to determine the degree of consistency of a microbiome-based classifier for each individual's salivary microbiome assessments (three total per subject).

CONTACTS AND LOCATIONS:
Overall Officials: Julian Abrams, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No